CLINICAL TRIAL: NCT04504838
Title: A Longitudinal, Observational Study to Explore the Tidal Breathing Carbon Dioxide (TBCO2) Waveform, Measured Using the N-Tidal C Device, in Asthma
Brief Title: The Asthma Breathing Record Study
Acronym: ABRS
Status: Completed | Type: Observational
Sponsor: TidalSense (Industry)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2019/26; 37872 (Other: ISRCTN)
Record Dates: First submitted 2020-04-08; First posted 2020-08-07 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study involves a new device, called 'N-Tidal C', which uses a method that has the potential to predict when asthma attacks are about to happen. The device works by accurately measuring an individual's exhaled CO2 waveform. A person has to breathe in and out through the mouthpiece at their normal relaxed rate of breathing. It does not need any extra effort and therefore has considerable benefits over current breathing tests which require significant patient effort.

DETAILED DESCRIPTION:
People with more severe asthma suffer from frequent asthma attacks that require regular hospital admissions. These attacks are difficult to predict and can devastate the lives of patients. A new tool is needed that can help to predict when an asthma attack is going to happen. This would help people recognise an attack earlier and allow treatment to be started sooner. This study will evaluate a new breathing monitor, to see whether it can detect asthma attacks. The study tests a new device, called 'N-Tidal C', which uses a method that has the potential to predict when attacks are about to happen. The investigators have found that people with asthma breathe out a gas, called carbon dioxide (CO2), in a different way to healthy people. The pattern of breathing out CO2 (the waveform) changes further when patients are having an attack of their disease. If patients could monitor their CO2, they may recognise when their asthma is getting worse, and take earlier action to avoid attacks getting out of hand and going to hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, aged ≥7 years.
2. Confirmed clinician diagnosis of asthma by examination of medical records, and based on accepted national and/or international criteria e.g. BTS/SIGN, or GINA.
3. Moderate or Severe asthma (defined as BTS stage 2-5)
4. Poorly controlled asthma (defined as an ACQ score of ≥1)
5. Exacerbation prone asthma (defined as at least 1 asthma exacerbation requiring oral corticosteroid treatment in the last 12 months).
6. Providing written informed consent, or parental/guardian consent and participant assent in the case of a child

Exclusion Criteria:

1. Inability to understand or comply with study procedures and/or inability to give fully informed consent.
2. Known other lung, chest wall, neuromuscular, cardiac or other comorbidity or abnormality that would affect spirometry and/or other measures of lung function or TBCO2 measurements (including Breathing Pattern Disorder or Chronic Obstructive Pulmonary Disease).
3. Smokers (current or ex-smokers) with a >10 pack year history.
4. In the opinion of the clinical investigator, the participant would have difficulty completing the study procedures consistently (for example, difficulty holding the device, or long periods of absence/travel) throughout the study period.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with poorly controlled asthma
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Tidal Breathing Carbon Dioxide (TBCO2) breath records measured by the N-Tidal C data collector device. | From baseline until study completion, up to 12 months.
  To collect Tidal Breathing Carbon Dioxide (TBCO2) breath records, twice daily per participant, which will be correlated to patient reported outcomes and clinical assessments.

SECONDARY OUTCOMES:
Disease Control in asthma patients | From baseline until study completion, up to 12 months.
  Asthma Control Questionnaire (ACQ) (0= no impairment 6 = maximum impairment)
Quality of Life | From baseline until study completion, up to 12 months.
  Asthma Quality of Life Questionnaire (AQLQ) 7 = not impaired at all - 1 = severely impaired
Usability and Acceptability of the device | From baseline until study completion, up to 12 months.
  Visual Analogue Scale (VAS) (7=easy to use - 28=difficult to use)
Impact on work activity of the device within asthma population | From baseline until study completion, up to 12 months.
  Work Productivity and Activity Impairment Questionnaire (WPAI): Asthma (1=employed - 5= health affected productivity while working)

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Chauhan, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Talker L, Neville D, Wiffen L, Selim AB, Haines M, Carter JC, Broomfield H, Lim RH, Lambert G; BRS Study Team; Weiss ST, Hayward G, Brown T, Chauhan A, Patel AX. Machine diagnosis of chronic obstructive pulmonary disease using a novel fast-response capnometer. Respir Res. 2023 Jun 2;24(1):150. doi: 10.1186/s12931-023-02460-z. PMID 37268935